CLINICAL TRIAL: NCT00880139
Title: A Cross-sectional Study Investigating the Levels and Effects of Low-grade Inflammation in Diabetic Retinopathy of Type 1 Diabetes
Brief Title: Study Investigating the Levels and Effects of Low-grade Inflammation in Diabetic Retinopathy of Type 1 Diabetes
Status: Terminated | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. - Doz. Dr, Medical University of Vienna
Other Study IDs: OPHT-171008
Record Dates: First submitted 2008-12-18; First posted 2009-04-13 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Diabetic Retinopathy; Inflammation
Keywords: Diabetes mellitus, type 1; Inflammation; Cytokines; Vascular reactivity
MeSH Terms: conditions — Diabetic Retinopathy; Inflammation; Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

INTERVENTIONS:
Procedure: Blood sampling — Determination of cytokine plasma levels (ELISA)
Procedure: Noninvasive measurement of systemic hemodynamics — performed once
Procedure: Visual acuity assessment — ETDRS charts
Device: Blue field entoptic technique (Blue field stimulator, BFS-2050) — performed once
  Other Names: Blue field stimulator; BFS-2050
Procedure: Ophthalmic examination and fundus photography — 7 + 1 standard fields
Device: Retinal Vessel Analyzer (DVA) — Assessment of retinal vessel reactivity to stimulation with flickering light
  Other Names: DVA
Device: High resolution optical coherence tomography (OCT) — performed once
  Other Names: OCT

SUMMARY:
There is much evidence that localized low grade inflammatory processes may contribute to the microvascular complications of type 1 and type 2 diabetes mellitus including sight-threatening diabetic retinopathy. Some biomarkers for inflammation have been found to be elevated in diabetes patients and correlations between those biomarkers and the severity of diabetic complications have been found in the last years. The relation between this low grade inflammation and the microvascular changes observed in diabetic retinopathy is, however, not well characterized.

In the present study patients with different stages of non-proliferative diabetic retinopathy will be included. Several markers of inflammation will be measured from blood samples. These markers will be related to vascular factors including flicker-induced vasodilatation as a marker of endothelial dysfunction and perifoveal leukocyte velocity and density as measured with the blue field entoptic phenomenon. In addition, the ophthalmologic status of the patients will be assessed according to the Modified Airlie House classification.

A multiple regression model will be employed to study the association between the different methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes mellitus with duration of > 1 year
* Men and women, age ≥ 18, nonsmokers
* Body mass index between 16 and 30 kg/m²
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant or diabetes-related
* Mild, moderate or severe non-proliferative diabetic retinopathy

Exclusion Criteria:

* Abuse of drugs or alcoholic beverages
* Participation in a clinical trial in the 3 weeks preceding the study
* Treatment with anti-inflammatory drugs in the 3 weeks before the study day
* Symptoms of a clinically relevant illness in the 3 weeks before the study day
* Blood donation or equivalent blood loss in the 3 weeks before the study day
* Other ocular pathologies than non-proliferative diabetic retinopathy
* Ametropia > 6 dpt
* History or family history of epilepsy
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Plasma biomarkers for inflammation (CRP, TNF-α, IL-6, vWF, e-Selektin) | 1 day
Perifoveal white cell blood flow (Blue field entoptic technique) | 1 day
Retinal vessel reactivity to flicker stimulation (Retinal Vessel Analyzer) | 1 day
Arteriolar to venous ratio | 1 day

SECONDARY OUTCOMES:
Capillary blood glucose | 1 day
Stage of diabetic retinopathy | 1 day
Visual acuity | 1 day
Intraocular pressure | 1 day
Systolic/diastolic arterial blood pressure, pulse rate | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Pemp, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria